CLINICAL TRIAL: NCT05026645
Title: Acute Care For Patients Exposed to a Chemical, Biological, Radiological, Nuclear, Explosive: Attack: Protocol For An International Multicentric Observational Study
Brief Title: The Medical Management in Patients Exposed to Weapons of Mass Destruction
Acronym: CBRNEObs
Status: Enrolling by invitation | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Quebec Heart and Lung Institute, Quebec City, Canada (Unknown); Sorbonne University (Other); Medical Intelligence CBRNE inc.; Quebec City, Canada (Unknown); Department of Intensive Care Medicine, Tokyo, Japan (Unknown); Centre for Defence and Security Studies, University of Manitoba, Winnipeg, Canada (Unknown); Biomedical Telematics Laboratory, Quebec Respiratory Health Research Network, Sherbrooke, Canada (Unknown); Tokyo University (Other); Tokyo Women's Medical University (Other); University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Stephane Bourassa, Chief of CBRNE Team, St. Justine's Hospital
Other Study IDs: 2020-2561
Record Dates: First submitted 2021-08-18; First posted 2021-08-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chemical Injury; Chemicals; Intoxication; Acute Respiratory Distress Syndrome; Distress Respiratory Syndrome; Medical Emergencies
Keywords: CBRNE Defence; Acute Settings; Pre-Hospital Settings; Decontamination; Protection; Respiratory Insults; Treatments
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Atelectasis | interventions — Decontamination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- adult inflicted by a CBRNE weapon: Part of the Population is being studied includes any individual who was affected by CBRNE attacks and needed an intervention of the healthcare system.
  Interventions: Procedure: Clinical interventions performed in acute settings (contaminated environment); Procedure: Protection (clinician and patient); Procedure: Decontamination (clinician and patient)
- Infant inflicted by a CBRNE weapon: Part of the population is being studied includes any individual who was affected by CBRNE attacks and needed an intervention of the healthcare system.
  Interventions: Procedure: Clinical interventions performed in acute settings (contaminated environment); Procedure: Protection (clinician and patient); Procedure: Decontamination (clinician and patient)
- Women inflicted by a CBRNE weapon: Part of the Population is being studied includes any individual who was affected by CBRNE attacks and needed an intervention of the healthcare system.
  Interventions: Procedure: Clinical interventions performed in acute settings (contaminated environment); Procedure: Protection (clinician and patient); Procedure: Decontamination (clinician and patient)
- Men inflicted by a CBRNE weapon: Part of the Population is being studied includes any individual who was affected by CBRNE attacks and needed an intervention of the healthcare system.
  Interventions: Procedure: Clinical interventions performed in acute settings (contaminated environment); Procedure: Protection (clinician and patient); Procedure: Decontamination (clinician and patient)
- Elderly inflicted by a CBRNE weapon: Part of the Population is being studied includes any individual who was affected by CBRNE attacks and needed an intervention of the healthcare system.
  Interventions: Procedure: Clinical interventions performed in acute settings (contaminated environment); Procedure: Protection (clinician and patient); Procedure: Decontamination (clinician and patient)
- Diagnosed with chronic disease(s) inflicted by a CBRNE weapon: Part of the Population is being studied includes any individual who was affected by CBRNE attacks and needed an intervention of the healthcare system.
  Interventions: Procedure: Clinical interventions performed in acute settings (contaminated environment); Procedure: Protection (clinician and patient); Procedure: Decontamination (clinician and patient)
- Clinician (adult) whom performs his/her clinical interventions: Clinician (adult) whom performs his/her clinical interventions while integrating competences in protections and decontamination. Part of the Population is being studied includes any individual who was affected by CBRNE attacks and needed an intervention of the healthcare system. This is the case of when the clinician is required to ensure safety toward his/her patient while performing his/her interventions & procedures.
  Interventions: Procedure: Clinical interventions performed in acute settings (contaminated environment); Procedure: Protection (clinician and patient); Procedure: Decontamination (clinician and patient)
- Clinician (adult) injured by duties circumstances: Part of the Population is being studied includes any individual who was affected by CBRNE attacks and needed an intervention of the healthcare system. This is the case of when the clinician becomes inflicted by a CBRNE weapon while intervening toward contaminated patient due to any failure in protection and decontamination.
  Interventions: Procedure: Clinical interventions performed in acute settings (contaminated environment); Procedure: Protection (clinician and patient); Procedure: Decontamination (clinician and patient)

INTERVENTIONS:
Procedure: Clinical interventions performed in acute settings (contaminated environment) — Any clinical intervention performed on the patient inflicted by at least one of Chemical, Biological, Radiological, Nuclear, Explosive (CBRNE) weapons in acute settings (from the incident site up to his/her admission to the clean zone of a emergency room or its equivalent (ie.: walking clinic).
Procedure: Protection (clinician and patient) — As interrelated competence of the clinical intervention, any protection procedure and capability applied on the patient inflicted by at least one of Chemical, Biological, Radiological, Nuclear, Explosive (CBRNE) weapons in acute settings (from the incident site up to his/her admission to the clean zone of a emergency room or its equivalent (ie.: walking clinic). Concerning the clinician, the protection implied for his/her own safety and for the patient to whom she/he was in closed/contact with.
Procedure: Decontamination (clinician and patient) — As interrelated competence of the clinical intervention and protection, any decontamination procedure and capability applied on the patient inflicted by at least one of Chemical, Biological, Radiological, Nuclear, Explosive (CBRNE) weapons in acute settings (from the incident site up to his/her admission to the clean zone of a emergency room or its equivalent (ie.: walking clinic). Concerning the clinician, the protection implied for his/her own safety and for the patient to whom she/he was in closed/contact with. This crucial step is usually expected prior the patient's transfer into a clean zone like the emergency room or its equivalent.

SUMMARY:
Observation study measuring medical response in contaminated environment.

DETAILED DESCRIPTION:
This is an ongoing multicentric observational study that aims to assess the medical response to chemical, biological, radiological, nuclear, explosive (cbrne) events during the last five (5) decades (i.e.: 1970-2020), and in any future cbrne attack that might occur within the next 15 years (i.e.: 2021-2036). Of note, the data collection will be performed retrospectively and after sites review ethic board (REB) approval.

ELIGIBILITY:
Inclusion Criteria:

i. a CBRNE attack caused at least one casualty who required the assistance of the participating health care system (e.g.: physicians, nurses, paramedics and other health-care specialists of a medical facility) during a medical extraction from the incident site until admission to a medical facility;

ii. Patients are eligible if they were exposed to the CBRNE attack;

iii. Medical information concerning the CBRNE exposures, even if partial, is accessible to health care professionals for the purposes of filling out the online case report form (eCRF);

iv. Participants must be able to complete the online case report form in English; and

v. The approval of an Ethics Review Board is obtained by each medical centre participant.

Exclusion Criteria:

A negative response to any of the inclusion criteria results in an exclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population is being studied includes any individual who was affected by CBRNE attacks and needed an intervention of the healthcare system.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2036-11-01 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
Intervention and location | At the patient's admission at the hospital emergency room (i.e.: end-point of the medical extraction/evacuation).
  The percentage of patients to whom the World Health Organization's healthcare guidelines were applied without any delay (i.e.: during a medical extraction/evacuation)

SECONDARY OUTCOMES:
Contamination is under-control due to efficient protective measures applied during a medical extraction/evacuation | At the patient's admission at the hospital emergency room (i.e.: end-point of the medical extraction/evacuation).
  The percentage of patients whose health condition remained stable during a medical extraction due to efficient WHO's protective measures applied
Contamination under-control due to efficient decontamination measures applied during a medical extraction/evacuation | At the patient's admission at the hospital emergency room (i.e.: end-point of the medical extraction/evacuation).
  The percentage of patients whose health condition remained stable during a medical extraction due to efficient WHO's decontamination measures applied
Deterioration of the patient's health condition due to compromised means of protection | At the patient's admission at the hospital emergency room (i.e.: end-point of the medical extraction/evacuation).
  The percentage of patients whose health condition deteriorate during a medical extraction due to the misuse of WHO's protective measures (e.g.: mask, suit, gloves, boots, etc).
Deterioration of the patient's health condition due to compromised means of decontamination | At the patient's admission at the hospital emergency room (i.e.: end-point of the medical extraction/evacuation).
  The percentage of patients whose health condition deteriorated during a medical extraction due to the misuse of WHO's decontamination measures (e.g.: immediate (roughly) or/and thorough (specialized one)).

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Bourassa, Principal Investigator — Ste-Justine's Hospital
Locations (15):
- Director, Unconventional Weapons & Technology Division, National Consortium for the Study of Terrorism and Responses to Terrorism University of Maryland, College Park, Maryland, United States
- Canada (7):
  - Centre for Defence and Security Studies, University of Manitoba, Winnipeg, Manitoba
  - Royal Canadian Medical Corps, Ottawa, Ontario
  - École de Technologie Supérieure Université du Québec, Montreal, Quebec
  - Research Center of the CHU St-Justine, University of Montreal, Montreal, Quebec
  - Research Centre, Quebec Heart and Lung Institute, Laval University, Québec, Quebec
  - Medical Intelligence CBRNE Inc., Québec, Quebec
  - Biomedical Telematics Laboratory Platform of the Quebec Respiratory Health Research Network, Sherbrooke, Quebec
- University of Finance and Administration Department of Criminology and Forensic Disciplines, Prague, Prague, Czechia
- Sorbonne University, Paris, Île-de-France Region, France
- Japan (3):
  - Tokyo Women's Medical University, Department of Intensive Care Medicine, Tokyo, Shinjuku-ku
  - Department of Critical care, Miyagi Children's Hospital, Tokyo
  - Department of Disaster Medical Management, The University of Tokyo Hospital, Tokyo
- United Kingdom (2):
  - Surrey and Sussex Healthcare NHS Trust, Surrey Quays, Redhill
  - CBRNE World Journal, Winchester

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, we do have any plan. However, for the interest of pursuing the research, that matter will require to be addressed in due time.

REFERENCES:
- [Derived] Bourassa S, Noebert D, Dauphin M, Rambaud J, Kawaguchi A, Leger F, Beijer D, Fortier Y, Dligui M, Ivanovski H, Simard S, Jouvet P, Leclerc J. Acute care for patients exposed to a chemical attack: protocol for an international multicentric observational study. BMJ Open. 2022 Sep 29;12(9):e065015. doi: 10.1136/bmjopen-2022-065015. PMID 36175098